CLINICAL TRIAL: NCT05788367
Title: Pericapsular Nerve Block Versus Interscalene Nerve Block for Acute Pain Management in Shoulder Arthroscopy: A Randomized Controlled Study
Brief Title: Pericapsular Nerve Block Versus Interscalene Nerve Block for Acute Pain Management in Shoulder Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Fouad Algyar, Lecturer of Anaesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Kafrelsheikh University, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MKSU 50-12-7
Record Dates: First submitted 2023-01-12; First posted 2023-03-28 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Pericapsular Nerve Block; Interscalene Nerve Block; Shoulder Arthroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The pericapsular nerve group (Active Comparator): patients received Ultrasound guided The pericapsular nerve group block using 20 ml of bupivacaine 0.5%
  Interventions: Procedure: The pericapsular nerve group
- Interscalene group (Active Comparator): patients will receive interscalene brachial plexus block using 15 ml of bupivacaine 0.5% before induction of general anesthesia.
  Interventions: Procedure: Interscalene brachial plexus block

INTERVENTIONS:
Procedure: The pericapsular nerve group — patients received Ultrasound guided pericapsular nerve group block using 20 ml of bupivacaine 0.5%
  Arms: The pericapsular nerve group
Procedure: Interscalene brachial plexus block — patients will receive interscalene brachial plexus block using 15 ml of bupivacaine 0.5% before induction of general anesthesia
  Arms: Interscalene group

SUMMARY:
The aim of this study is to compare PENG and ISB after shoulder arthroscopy for postoperative pain management after shoulder arthroscopy.

DETAILED DESCRIPTION:
Shoulder arthroscopy is a common procedure done is orthopedics for many surgical indications as rotator cuff tears, stiffness and instability. This procedure has a well - documented postoperative pain. To improve the outcome after surgery, effective pain control is needed.

Various methods are used for postoperative pain management. Intravenous opioid agents are among them, but they may cause undesirable side effects, such as respiratory depression, sedation, constipation, allergic reaction, nausea, and vomiting. Thus, alternative techniques are preferred.

Interscalene brachial plexus blocks (ISBPBs) are often used to provide perioperative analgesia and anesthesia for shoulder surgery. They target nerve roots C4-C6 and thereby provide regional analgesia to the shoulder and upper arm. Although ISBPBs are often performed in combination with general anesthesia (GA) to enhance postoperative analgesia, they are also sometimes used as a sole means of anesthesia.

The pericapsular nerve group (PENG) block is an ultrasound-guided approach, first described by Giron-Arango et al. for the blockade of the articular branches of the femoral, obturator and accessory obturator nerves that provide sensory innervation to the anterior hip capsule. It has been successfully used as an alternative regional anaesthesia technique for the management of acute pain after hip fracture, and for analgesia after elective hip surgery

ELIGIBILITY:
Inclusion Criteria:

* Body mass index < 40 kg/m2
* American Society of Anesthesiologists (ASA) physical status I-II
* posted for elective shoulder arthroscopy

Exclusion Criteria:

* Known allergy to local anesthetics
* allergy to all opioid medications
* diagnostic shoulder arthroscopic procedures
* patients with chronic opioids use and coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-10-05 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Asses The postoperative opioid consumption | 24 hours postoperatively
  the postoperative opioid consumption during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed F Algyar, MD, Principal Investigator — Lecturer of Anaesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Kafrelsheikh University
Locations (1):
- Mohammed Fouad Mohamed Algyar, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be provided under a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after the end of the study